CLINICAL TRIAL: NCT06260527
Title: A Phase 1, Randomized, Double-blind, Third-party Open, Placebo-controlled Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Food Effect After Single and Multiple Oral Doses of ARTS-011 In Chinese Health Subjects
Brief Title: Safety and Pharmacokinetic Study of ARTS-011 in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allorion Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ARTS-011-101
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Chinese Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: Single ascending dose (SAD) following by multiple ascending dose (MAD) and food effect study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single ascending dose (SAD) (Experimental): ARTS-011 and placebo will be randomized assigned and single dose administrated.
  Interventions: Drug: ARTS-011; Drug: Placebo
- Multiple ascending dose (MAD) (Experimental): ARTS-011 and Placebo will be randomized assigned and continuously administrated once daily for 7 days.
  Interventions: Drug: ARTS-011; Drug: Placebo
- Food effect study (Experimental): ARTS-011 will be single administered under the fasting and high-fat meal condition.
  Interventions: Drug: ARTS-011

INTERVENTIONS:
Drug: ARTS-011 — Single ascending dose (SAD): 3mg, 10mg, 20mg, 40mg, and 60mg. Multiple ascending dose (MAD): 10mg QD, 20mg QD, and 40mg QD X 7 days. Food effect study: single dose of ARTS-011 under the fasting and high-fat meal.
Drug: Placebo — Multiple ascending dose (MAD): 10mg QD, 20mg QD, and 40mg QD X 7 days. Multiple ascending dose (MAD): 10mg QD, 20mg QD, and 40mg QD X 7 days.
  Arms: Multiple ascending dose (MAD); Single ascending dose (SAD)

SUMMARY:
This single- and multiple-ascending dose study is a Phase 1, first in human study of ARTS-011. The goal of the study is to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of ARTS-011 after single and multiple oral doses of ARTS-011 in Chinese healthy volunteers.

DETAILED DESCRIPTION:
ARTS-011 is an oral potent Tyrosine kinase 2 (TYK2) inhibitor with a good selectivity profile over other human kinase. TYK2 is required for signal transduction and cellular functions downstream of interferons (IFN), IL-23, and IL-12 which are involved in the initiation and pathogenesis of psoriatic diseases. ARTS-011 is being developed for treatment of moderate-severe psoriasis and other autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male subjects between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 19.0 to 28.0 kg/m2; and a total body weight male ≥50.0 kg, female ≥45.0 kg.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* No evidence or history of clinically significant abnormalities of , vital signs (body temperature, pulse and blood pressure), laboratory tests (blood hematology and biochemistry, urine and coagulation function), 12-lead ECG and other examinations.
* Subjects has no fertility and sperm donation, egg donation plan and takes highly effective contraception during correctly for the duration of the active treatment period and for at least 90 days after the last dose of investigational drugs.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 150 mL) of wine or 360 mL of beer or 45 mL of hard liquor within 3 months of screening.
* History of tobacco/nicotine containing products in excess of >5 cigarettes/day within 3 months of screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product, whichever is longer.
* 12-lead ECG demonstrating QTc >450, or a QRS interval >120 msec at Screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc (or QRS) values should be used to determine the subject's eligibility.
* Screening laboratory abnormalities as defined by the protocol.
* Unwilling or unable to comply with the Lifestyle Guidelines as defined by the protocol.
* Subjected is not appropriate to be enrolled in the study per investigator's assessment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Discontinuation Due to AEs | SAD Cohort: Baseline up to Day 8, MAD Cohort: Baseline up to Day 14, Food Effect Cohort: Baseline up to Day 15
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
  An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug up to the end of study that are absent before treatment or that worsened relative to pretreatment state.
Number of Adverse Events (AEs) according to severity | SAD Cohort: Baseline up to Day 8, MAD Cohort: Baseline up to Day 14, Food Effect Cohort: Baseline up to Day 15
  AEs are classified according to the severity in 3 categories:
  1. mild - AEs does not interfere with participant's usual function
  2. moderate - AEs interferes to some extent with participant's usual function
  3. severe - AEs interferes significantly with participant's usual function
Number of participants with change from baseline in vital signs (blood pressure, pulse rate, oral temperature) | SAD Cohort: Baseline up to Day 8, MAD Cohort: Baseline up to Day 14, Food Effect Cohort: Baseline up to Day 15
Number of participants with change from baseline in 12-Lead Parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) | SAD Cohort: Baseline up to Day 8, MAD Cohort: Baseline up to Day 14, Food Effect Cohort: Baseline up to Day 15
  Electrocardiogram (ECG)
Number of participants with change from baseline physical examination | SAD Cohort: Baseline up to Day 8, MAD Cohort: Baseline up to Day 14, Food Effect Cohort: Baseline up to Day 15
  Physical examinations included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems.
Incidence and magnitude of treatment emergent clinical laboratory abnormalities | SAD Cohort: Baseline up to Day 8, MAD Cohort: Baseline up to Day 14, Food Effect Cohort: Baseline up to Day 15
  Criteria for abnormalities:
  Hematology: hemoglobin, hematocrit, red blood cell count: less than(<) 0.8*lower limit of normal (LLN); platelets: <0.5*LLN or >1.75*ULN, white blood cell count: <0.6*LLN or >1.5*ULN; lymphocytes, total neutrophils: <0.8*LLN or >1.2*ULN; eosinophils, basophils, monocytes: >1.2*ULN;
  Coagulation: activated partial thromboplastin time, prothrombin, prothrombin international ratio: >1.1*ULN;
  Liver function: bilirubin: >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >3.0*ULN; protein, albumin: <0.8*LLN></0>1.2*ULN;
  Renal function: blood urea nitrogen, creatinine: >1.3*ULN; uric acid: >1.2*ULN;
  Chemistry: sodium, potassium, chloride, calcium, bicarbonate: <0.9*LLN, or >1.1*ULN;
  Fasting glucose: <0.6*LLN, or >1.5*ULN;
  Urinalysis: pH<4.5, or >8; glucose, protein, blood, ketones, urobilinogen, bilirubin, nitrite.
Number of participants with change in 24-hour creatine clearance from baseline | SAD Cohort: Baseline and Day 1, MAD Cohort: Baseline and Day 7
  Creatinine clearance is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ARTS-011 in Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) | SAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose on Day 1; MAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 7
Time to Reach Maximum Observed Plasma Concentration (Tmax) of ARTS-011 in Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) | SAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose on Day 1; MAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 7
Dose Normalized Maximum Observed Plasma Concentration (Cmax[dn]) of ARTS-011 in Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) | SAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose on Day 1; MAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 7
  Dose normalized (dn) Cmax is calculated by dividing Cmax by the exact dose of ARTS-011 (in mg) administered to a participant.
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) of ARTS-011 in Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) | SAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose on Day 1; MAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 7
Plasma Decay Half-Life (t1/2) of ARTS-011 in Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) | SAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose on Day 1; MAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 7
Apparent Volume of Distribution (Vz/F) of ARTS-011 in Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) | SAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose on Day 1; MAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 7
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Apparent Clearance (CL/F) of ARTS-011 in Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) if data permit | SAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose on Day 1; MAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 7
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Clearance obtained after oral dose is influenced by the fraction of the dose absorbed. CL/F =Dose of ARTS-011/AUCinf.
Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of ARTS-011 in Single Ascending Dose (SAD) | SAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose on Day 1
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of ARTS-011 in Multiple Ascending Dose (MAD) | MAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 7
  Area under the plasma concentration versus time curve from time 0 to end of dosing interval (AUCtau), where dosing interval is 24 hours for MAD once daily.
Dose Normalized Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf[dn]) of ARTS-011 in Single Ascending Dose (SAD) | SAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose on Day 1
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). AUCinf(dn) was calculated by dividing AUCinf by the exact dose of ARTS-011 (in mg) administered to a participant.
Dose Normalized Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau[dn]) of ARTS-011 in Multiple Ascending Dose (MAD) | MAD: predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 7
  Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval is 24 hours for MAD once daily. AUCtau(dn) is calculated by dividing AUCtau by the exact dose of of ARTS-011 (in mg) administered to a participant.
Maximum Observed Plasma Concentration (Cmax) of ARTS-011 in Food Effect Cohort | Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 8
Time to Reach Maximum Observed Plasma Concentration (Tmax) of ARTS-011 in Food Effect Cohort | Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 8
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) of ARTS-011 in Food Effect Cohort | Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 8
Plasma Decay Half-Life (t1/2) of ARTS-011 in Food Effect Cohort | Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 8
Apparent Clearance (CL/F) of ARTS-011 in Food Effect Cohort if data permit | Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 8
Apparent Volume of Distribution (Vz/F) of ARTS-011 in Food Effect Cohort if data permit | Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose on Day 1 and Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Dong, MD, Principal Investigator — Beijing Friendship Hospital, Capital Medical University, China
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No